CLINICAL TRIAL: NCT00895414
Title: The Effect of Enalapril on Doxorubicin Exposure in Adjuvant Breast Cancer Treatment
Brief Title: Enalapril Maleate and Doxorubicin Hydrochloride in Treating Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008NTLS060; 0806M34981 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Enalapril; Enalaprilat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxorubicin alone first, then Doxorubicin with Enalapril (Experimental): Patients receive doxorubicin hydrochloride IV over 5-10 minutes on day 1. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 week before course 2, patients also receive oral enalapril maleate once daily until day 8 of course 2.
  Interventions: Drug: doxorubicin hydrochloride; Drug: enalapril maleate
- Doxorubicin with Enalapril first, then Doxorubicin alone (Experimental): Patients receive doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 week before course 1, patients receive oral enalapril maleate once daily until day 8 of course 1.
  Interventions: Drug: doxorubicin hydrochloride; Drug: enalapril maleate

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV 5-10 minutes on day 1. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Adriamycin
Drug: enalapril maleate — Given orally - Beginning 1 week before course 2, patients also receive oral enalapril maleate once daily until day 8 of course 2. OR Beginning 1 week before course 1, patients receive oral enalapril maleate once daily until day 8 of course 1.
  Other Names: Vasotec

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Enalapril maleate may help protect heart cells from the side effects of chemotherapy. It is not yet known whether giving enalapril maleate before or after doxorubicin hydrochloride is more effective in treating women with breast cancer.

PURPOSE: This randomized clinical trial is studying giving enalapril maleate together with doxorubicin hydrochloride to see how well it works in treating women with breast cancer.

DETAILED DESCRIPTION:
This study is a drug interaction study designed to study the effects of enalapril on doxorubicin metabolism. Women with breast cancer for whom at least two cycles every 14 day doxorubicin is planned will be considered for enrollment. Study participation will be for 2 treatment cycles of doxorubicin or approximately 4 weeks. Patients will receive a 14 day course of daily enalapril in association with one cycle of doxorubicin and receive no study agent during the other cycle allowing patients to act as their own control. The sequence of enalapril dosing will be assigned by randomization at study enrollment. Blood samples for pharmacokinetics will be drawn before and at 7 time points after each of the two doses of doxorubicin. For each patient, serum doxorubicin and doxorubicinol concentrations both on and off of enalapril will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Tissue diagnosis of a breast carcinoma
* The oncologist must have prescribed doxorubicin as part of the planned chemotherapy regimen
* Have acceptable organ function within 14 days of enrollment defined as:

  * liver function: total bilirubin, AST and ALT within normal institutional limits
  * kidney function: estimated Creatinine Clearance > 60 ml/min calculated creatinine clearance (for females) - formula: (140 - age) x weight x .85 divided by (sCr x 72)
* At least 18 years old
* Patient must have given written informed consent indicating an understanding of the investigational nature of the study
* Agrees not to consume grapefruit juice while on the study

Exclusion Criteria:

* Known allergy to enalapril
* Taking any known P450 cytochrome inducers or inhibitors
* Taking any herbal supplements while on the study or the week prior to receiving doxorubicin
* Taking an ace-inhibitor or angiotensin receptor blocker
* Pregnant or lactating. Enalapril is Pregnancy Categories C (first trimester) and D (second and third trimesters)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-04; Primary Completion 2014-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne H. Blaes, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Fairview Southdale Hospital, Edina, Minnesota
  - University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxorubicin Alone First, Then Doxorubicin With Enalapril: Patients receive doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Beginning 1 week before course 2, patients additionally receive oral enalapril maleate once daily until day 8 of course 2.
- Doxorubicin With Enalapril First, Then Doxorubicin Alone: Patients receive doxorubicin hydrochloride IV on day 1. Treatment repeats every 14 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Beginning 1 week before course 1, patients additionally receive oral enalapril maleate once daily until day 8 of course 1.
Period: First Intervention (14 Days)
Arm/Group | Doxorubicin Alone First, Then Doxorubicin With Enalapril | Doxorubicin With Enalapril First, Then Doxorubicin Alone
Started | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Second Intervention (14 Days)
Arm/Group | Doxorubicin Alone First, Then Doxorubicin With Enalapril | Doxorubicin With Enalapril First, Then Doxorubicin Alone
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients who were randomized to receive either doxorubicin hydrochloride alone or doxorubicin hydrochloride with enalapril.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Doxorubicin Plasma Concentrations Demonstrating a Significant Increase or Decrease When Doxorubicin Was Given With Enalapril as Compared to When Doxorubicin Was Given Without Enalapril.
Description: Doxorubicin plasma concentration (DPC) is the primary pharmacokinetic (PK) measure of the exposure. Each patient will have serial PKs performed twice - once with enalapril and once without enalapril. A mean increase or decrease of more than 115 ng/ml in DPC will be considered significant.
Time Frame: Baseline, 0.5, 1.0, 2.0, 4.0, 24.0 and 48.0 hours after infusion of doxorubicin
Measure: Number; unit: participants
Groups:
- Doxorubicin Hydrochloride Alone: Participants who received doxorubicin hydrochloride alone in either Cycle 1 or Cycle 2.
- Doxorubicin Hydrochloride With Enalapril: Participants who received doxorubicin hydrochloride with enalapril in either Cycle 1 or Cycle 2.
Arm/Group | Doxorubicin Hydrochloride Alone | Doxorubicin Hydrochloride With Enalapril
Number analyzed (Participants) | 17 | 17
participants | 0 | 0

2. Secondary Outcome: The Number of Participants With a Significant Increase or Decrease in the Baseline Levels of Btype Natriuretic Peptide, Cardiac Troponins, and Urine Microalbumin With or Without Enalapril
Description: Doxorubicin can induce changes in troponin, b-type natriuretic peptide and urine microalbumin. This analysis will determine whether enalapril prevents any of these changes. Statistical significance defined as a p < 0.05.
Time Frame: Baseline, 4, 24 and 48 hours after infusion of doxorubicin
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Hydrochloride Alone | Doxorubicin Hydrochloride With Enalapril
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

3. Secondary Outcome: The Number of Participants With a Significant Increase or Decrease in Doxorubicin Hydrochloride Metabolite Levels With or Without Enalapril
Description: Doxorubicin is metabolized to doxorubicinol. The effects of enalapril on doxorubicinol will be assessed. Statistical significance defined as a p < 0.05.
Time Frame: Baseline, 0.5, 1.0, 2.0, 4.0, 24.0 and 48.0 hours after infusion of doxorubicin
Measure: Count of Participants; unit: Participants
Arm/Group | Doxorubicin Hydrochloride Alone | Doxorubicin Hydrochloride With Enalapril
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Description: The adverse events could not be reported per intervention because the arms themselves were designed originally as one being "Doxorubicin Alone First, Then Doxorubicin With Enalapril" and the other being "Doxorubicin With Enalapril First, Then Doxorubicin Alone." As such the data was collected and reported under these two arms and it would not be possible further separate the adverse events by "Doxorubicin Hydrochloride Alone" and "Doxorubicin Hydrochloride With Enalapril."
Arm/Group | Doxorubicin Alone First, Then Doxorubicin With Enalapril | Doxorubicin With Enalapril First, Then Doxorubicin Alone
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 3/8 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin Alone First, Then Doxorubicin With Enalapril (N=8) | Doxorubicin With Enalapril First, Then Doxorubicin Alone (N=9)
tingling (Nervous system disorders) | 0 | 1
lightheaded (Nervous system disorders) | 0 | 1
dizziness (Nervous system disorders) | 3 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
headache (Nervous system disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1
chest pain, NOS (Gastrointestinal disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
palpitations (Cardiac disorders) | 1 | 0
food poisoning (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes